CLINICAL TRIAL: NCT01612676
Title: An Open Label Feasibility Trial Investigating FE 202158 as Potential Primary Vasopressor Treatment in Patients With Vasodilatory Hypotension in Early Septic Shock.
Brief Title: Investigating FE 202158 as Potential Primary Treatment in Patients With Early Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000025; 2012-001254-26 (EudraCT Number)
Record Dates: First submitted 2012-05-11; First posted 2012-06-06 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — vasopressin, Phe(2)-Ile(3)-Hgn(4)-Orn(iPr)(8)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug (Experimental): FE 202158
  Interventions: Drug: FE 202158

INTERVENTIONS:
Drug: FE 202158

SUMMARY:
The purpose of this trial is to investigate the potential of FE 202158 as a treatment which can stabilize blood pressure for treatment of patients in early septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form by the patient or a legal representative according to local regulations'
* Man or women 18 years of age or older
* Body weight below 115 kg for male patients and 100 kg for female patients
* Proven or suspected infection
* Septic shock, i.e. vasodilatory hypotension requiring vasopressor support
* Willing to use an adequate barrier method or hormonal method of contraception, if not abstinent, from informed consent to one week after the end of infusion of study medication

Exclusion Criteria:

* Present or a history within the last 6 months of symptoms of acute coronary syndrome (myocardial infarction or unstable angina)
* Known or suspected endocarditis
* Hypovolaemia suspected on clinical grounds, e.g. cold extremities with delayed capillary filling, low cardiac filling pressure, marked systolic or pulse pressure variation or positive leg raising test
* Known or suspected cardiac failure
* Known or suspected infection with (HIV)-1, HIV-2, hepatitis B, or hepatitis C
* Pregnancy or breastfeeding
* Any cause of hypotension other than early septic shock
* Use of vasopressin or terlipressin within 7 days prior to start of IMP infusion
* Proven or suspected acute mesenteric ischemia, as judged by the investigator
* Known episode of septic shock within 1 month prior to screening
* Death anticipated within 24 hours, or due to the underlying disease within 3 months
* Known past or current 2nd and 3rd degree AV-block without a well functioning pacemaker
* Brain injury within current hospitalisation
* Present hospitalisation with burn injury
* Symptomatic peripheral vascular disease including Raynaud's syndrome
* Previously included in this trial
* Intake of an Investigational Medicinal Product (IMP) within the last 3 months (or longer if judged by the Investigator to possibly influence the outcome of the current study)
* Known participation in another interventional clinical trial
* Considered by the investigator to be unsuitable to participate in the trial for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (4):
- Belgium (3):
  - Erasme Hospital Free University of Brussels, Brussels
  - Saint-Luc University Hospital, Brussels
  - University Hospital Brussels, Brussels
- Hvidovre Hospital, Hvidovre, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited at the respective intensive care units at four centers (3 in Belgium and 1 in Denmark) between 05 Jul 2012 to 15 Nov 2013.
Pre-assignment Details: Of the 159 patients screened, 31 patients were randomised and 30 patients were dosed. One patient in the 3.75 ng/kg/min dose group did not receive any study treatment due to an adverse event (elevation of troponin) recorded prior to infusion.
Groups:
- Infusion Regimen 1: 3.75 ng/kg/Min: FE 202158 0.1 mg/mL (10 mM acetate buffer, pH 4) was administered at initial infusion rate of 2.5 ng/kg/min, adjustable up to 3.75 ng/kg/min. Each patient received FE 202158 until recovered from the shock, however for not more than 7 days.
- Infusion Regimen 2: 5.0 ng/kg/Min: FE 202158 0.1 mg/mL (10 mM acetate buffer, pH 4) was administered at initial infusion rate of 2.5 ng/kg/min, adjustable up to 5.0 ng/kg/min. Each patient received FE 202158 until recovered from the shock, however for not more than 7 days.
- Infusion Regimen 3: 7.5 ng/kg/Min: FE 202158 0.1 mg/mL (10 mM acetate buffer, pH 4) was administered at initial infusion rate of 2.5-3.75 ng/kg/min adjustable up to a maximum of 7.5 ng/kg/min. Each patient received FE 202158 until recovered from the shock, however for not more than 7 days.
- Infusion Regimen 4: Modified 3.75 ng/kg/Min: FE 202158 0.1 mg/mL (10 mM acetate buffer, pH 4) was administered at initial infusion rate of 2.5-3.75 ng/kg/min, allowed to be increased to a maximum of 7.5 ng/kg/min if needed, with a maximum duration of 1 hour, during the first 6 hours of infusion. After 1 hour, or beyond the initial 6 hours, the infusion rate could not exceed 3.75 ng/kg/min. Each patient received FE 202158 until recovered from the shock, however for not more than 7 days.
Period: Overall Study
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Started | 6 | 7 | 5 | 13
Dosed | 5 | 7 | 5 | 13
Completed | 4 | 3 | 4 | 10
Not Completed | 2 | 4 | 1 | 3
Not completed — Adverse Event | 2 | 3 | 1 | 3
Not completed — Protocol Violation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Groups:
- Infusion Regimen 1: FE 202158 0.1 mg/ml (10 mM acetate buffer, pH 4) was administered at initial infusion rate of 2.5 ng/kg/min, adjustable up to 3.75 ng/kg/min. Each patient received FE 202158 until recovered from the shock, however for not more than 7 days.
- Infusion Regimen 2: FE 202158 0.1 mg/ml (10 mM acetate buffer, pH 4) was administered at initial infusion rate of 2.5 ng/kg/min, adjustable up to 5.0 ng/kg/min. Each patient received FE 202158 until recovered from the shock, however for not more than 7 days.
- Infusion Regimen 3: FE 202158 0.1 mg/ml (10 mM acetate buffer, pH 4) was administered at initial infusion rate of 2.5-3.75 ng/kg/min adjustable up to a maximum of 7.5 ng/kg/min. Each patient received FE 202158 until recovered from the shock, however for not more than 7 days.
- Infusion Regimen 4: FE 202158 0.1 mg/ml (10 mM acetate buffer, pH 4) was administered at initial infusion rate of 2.5-3.75 ng/kg/min, allowed to be increased to a maximum of 7.5 ng/kg/min if needed, with a maximum duration of 1 hour, during the first 6 hours of infusion. After 1 hour, or beyond the initial 6 hours, the infusion rate could not exceed 3.75 ng/kg/min. Each patient received FE 202158 until recovered from the shock, however for not more than 7 days.
- Total: Total of all reporting groups
Arm/Group | Infusion Regimen 1 | Infusion Regimen 2 | Infusion Regimen 3 | Infusion Regimen 4 | Total
Number analyzed (Participants) | 5 | 7 | 5 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (12.7) | 67.9 (13.7) | 64.8 (10.1) | 67.6 (13.2) | 67.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5 | 10
  Male | 4 | 5 | 3 | 8 | 20
Weight [Mean (Standard Deviation); unit: kg] | 66.6 (13.5) | 74.7 (17.7) | 81.3 (8.0) | 78.9 (15.3) | 76.3 (14.8)
Total Sequential Organ Failure Assessment Score [Mean (Standard Deviation); unit: Score on scale] — The Sequential Organ Failure Assessment score (SOFA) score is a scoring system to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems.
  The total SOFA score is a sum of the individual scores and range from 4 to 24, 4 being the best and 24 being the worst patient status.
  Score on scale | 11 (3.32) | 10 (2.31) | 8.8 (3.19) | 9.31 (3.01) | 9.67 (2.88)
Septic shock characteristic: Primary infection type [Number; unit: patients]
  Bacterial | 4 | 6 | 3 | 12 | 25
  Unknown | 0 | 1 | 1 | 1 | 3
  Other | 1 | 0 | 1 | 0 | 2
Septic shock characteristic: Primary infection location [Number; unit: patients]
  Abdominal cavity | 1 | 5 | 3 | 6 | 15
  Lung | 1 | 1 | 0 | 1 | 3
  Urinary tract | 0 | 1 | 1 | 4 | 6
  Other | 3 | 0 | 1 | 1 | 5
  Unknown | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Maintaining Target/Adequate Mean Arterial Pressure (MAP>60 mmHg) Without Norepinephrine
Description: Mean arterial pressure (MAP) was measured intra-arterially on a continuous basis. Success percentage of patients maintaining target/adequate MAP (>60 mmHg) without norepinephrine is presented.
Time Frame: Day 1 up to Day 7 post-infusion (Data collected at Day 1 at 1, 2, 3, 4, 5, 6, 9, 12, 15, 18 and 24 h, Day 2 at 36 and 48 h, Day 3 at 72 h, Day 4 at 96 h, Day 5 at 120 h, Day 6 at 144 h, and Day 7 at 168 h). Data is presented for specific time points.
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Measure: Number (60% Confidence Interval); unit: Percentage of patients
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 5 | 13
Percentage of patients
  Day 1 (Post 1 h) | 20.0 [4.4 to 49.0] | 42.9 [22.8 to 65.0] | 60.0 [32.7 to 83.1] | 7.7 [1.7 to 21.3]
  Day 1 (Post 3 h) | 20.0 [4.4 to 49.0] | 14.3 [3.1 to 37.1] | 60.0 [32.7 to 83.1] | 53.8 [38.7 to 68.4]
  Day 1 (Post 6 h) | 25.0 [5.4 to 58.2] | 14.3 [3.1 to 37.1] | 80.0 [51.0 to 95.6] | 76.9 [61.6 to 88.0]
  Day 1 (Post 12 h) | 60.0 [32.7 to 83.1] | 28.6 [12.0 to 51.7] | 80.0 [51.0 to 95.6] | 53.8 [38.7 to 68.4]
  Day 1 (Post 18 h) | 60.0 [32.7 to 83.1] | 42.9 [22.8 to 65.0] | 80.0 [51.0 to 95.6] | 66.7 [50.3 to 80.2]
  Day 1 (Post 24 h) | 80.0 [51.0 to 95.6] | 42.9 [22.8 to 65.0] | 80.0 [51.0 to 95.6] | 61.5 [46.1 to 75.2]
  Day 2 (Post 36 h) | 80.0 [51.0 to 95.6] | 66.7 [41.5 to 86.0] | 80.0 [51.0 to 95.6] | 61.5 [46.1 to 75.2]
  Day 2 (Post 48 h) | 80.0 [51.0 to 95.6] | 50.0 [26.9 to 73.1] | 80.0 [51.0 to 95.6] | 76.9 [61.6 to 88.0]
  Day 3 (Post 72 h) | 80.0 [51.0 to 95.6] | 66.7 [41.5 to 86.0] | 80.0 [51.0 to 95.6] | 69.2 [53.7 to 81.8]
  Day 4 (Post 96 h) | 80.0 [51.0 to 95.6] | 80.0 [51.0 to 95.6] | 80.0 [51.0 to 95.6] | 76.9 [61.6 to 88.0]
  Day 5 (Post 120 h) | 80.0 [51.0 to 95.6] | 80.0 [51.0 to 95.6] | 80.0 [51.0 to 95.6] | 84.6 [69.9 to 93.6]
  Day 6 (Post 144 h) | 80.0 [51.0 to 95.6] | 80.0 [51.0 to 95.6] | 80.0 [51.0 to 95.6] | 84.6 [69.9 to 93.6]
  Day 7 (Post 168 h) | 80.0 [51.0 to 95.6] | 80.0 [51.0 to 95.6] | 80.0 [51.0 to 95.6] | 76.9 [61.6 to 88.0]

2. Secondary Outcome: Urinary Output
Description: The urinary output was recorded every 24 hours up to Day 7, or as long as the patient was in intensive care unit.
Time Frame: Day 1 up to Day 7 post-infusion (Data collected on Day 1 at 24 h, Day 2 at 48 h, Day 3 at 72 h, Day 4 at 96 h, Day 5 at 120 h, Day 6 at 144 h, and Day 7 at 168 h). Data is presented for specific time points.
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Measure: Mean (60% Confidence Interval); unit: mL/kg
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 5 | 13
mL/kg
  Day 1 (Post 24 h) | 24.9 [16.0 to 33.8] | 21.8 [16.4 to 27.2] | 36.0 [27.0 to 45.1] | 24.1 [20.2 to 28.0]
  Day 2 (Post 48 h) | 42.9 [26.7 to 59.1] | 31.0 [23.9 to 38.0] | 55.9 [41.8 to 69.9] | 48.1 [36.6 to 59.5]
  Day 3 (Post 72 h) | 57.3 [32.3 to 82.3] | 43.2 [32.3 to 54.1] | 79.2 [58.0 to 100.4] | 72.3 [53.7 to 91.0]
  Day 4 (Post 96 h) | 68.0 [37.6 to 98.4] | 58.8 [42.1 to 75.4] | 100.5 [74.4 to 126.7] | 94.0 [69.4 to 118.7]
  Day 5 (Post 120 h) | 74.3 [42.3 to 106.3] | 73.3 [51.1 to 95.6] | 125.2 [94.3 to 156.1] | 106.2 [79.2 to 133.2]
  Day 6 (Post 144 h) | 81.8 [46.6 to 116.9] | 85.9 [58.2 to 113.5] | 139.8 [104.7 to 175.0] | 111.9 [84.8 to 139.1]
  Day 7 (Post 168 h) | 82.0 [46.8 to 117.2] | 96.1 [64.2 to 128.0] | 144.7 [108.2 to 181.2] | 115.1 [87.7 to 142.5]

3. Secondary Outcome: Fluid Balance
Description: The fluid balance (accumulated input/output) was recorded in 24-hour collecting periods when the patient was in the intensive care unit and during the infusion of FE 202158.
Time Frame: as for outcome 2
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Measure: Mean (60% Confidence Interval); unit: mL/kg
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 5 | 13
mL/kg
  Day 1 (Post 24 h) | 50 [23 to 77] | 72 [60 to 85] | 62 [50 to 74] | 61 [52 to 69]
  Day 2 (Post 48 h) | 69 [34 to 103] | 128 [103 to 153] | 96 [78 to 113] | 75 [66 to 85]
  Day 3 (Post 72 h) | 75 [32 to 118] | 173 [141 to 206] | 115 [94 to 135] | 72 [61 to 83]
  Day 4 (Post 96 h) | 76 [30 to 122] | 189 [153 to 226] | 107 [90 to 124] | 68 [57 to 79]
  Day 5 (Post 120 h) | 80 [31 to 130] | 209 [172 to 247] | 90 [78 to 102] | 69 [57 to 81]
  Day 6 (Post 144 h) | 84 [31 to 138] | 209 [166 to 252] | 88 [75 to 100] | 76 [61 to 91]
  Day 7 (Post 168 h) | 90 [33 to 147] | 220 [174 to 267] | 98 [77 to 119] | 78 [62 to 95]

4. Secondary Outcome: Summary of Investigator Reported Outcomes
Description: Investigator reported outcome on FE 202158 performance. Answers were graded on a visual analogue scale (VAS) from 0 to 10, 0 being the worst and 10 being the best outcome.
Time Frame: Day 1 up to Day 2
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 5 | 13
Score on scale
  Onset of action adequate to reach target MAP | 4.4 (3.78) | 3.57 (2.51) | 9.0 (1.22) | 7.85 (2.54)
  MAP maintained within desired boundaries (Day 1) | 6.8 (2.77) | 3.86 (2.67) | 9 (1.22) | 7.69 (3.66)
  MAP maintained within desired boundaries (Day 2) | 10 (0) | 4 (2.35) | 8.75 (1.26) | 6.71 (3.77)
  Confidence to use FE 202158 as primary treatment | 6.5 (1.91) | 5.5 (2.43) | 9.5 (0.577) | 8.18 (2.44)

5. Secondary Outcome: Morbidity Assessment
Description: Percentage of all the "Days alive and out/free of" intensive care unit, hospital, dialysis, or ventilation within Day 28 were summarized. Patients dying before or at Day 28 were counted as zero.
Time Frame: Day 1 up to Day 28
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Measure: Number; unit: percentage of days within 28 days
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 5 | 13
percentage of days within 28 days
  Days alive and out of intensive care unit | 51.6 | 31.4 | 61.2 | 58.8
  Days alive and out of hospital | 12.8 | 3.6 | 17.8 | 26.2
  Days alive and free of dialysis | 60 | 38.6 | 80 | 76.7
  Days alive and free of ventilation | 58.8 | 39.6 | 75.6 | 73.9

6. Secondary Outcome: Graded Morbidity
Description: Collection of data on graded morbidity was performed on Day 28 in addition to the collection of data on time of stay in intensive care unit and hospital.
Time Frame: Day 1 up to Day 28
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Measure: Number; unit: patients
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 5 | 13
patients
  Alive and out of hospital | 2 | 0 | 2 | 6
  In hospital (not intensive care unit) | 1 | 2 | 2 | 4
  In intensive care unit | 1 | 1 | 0 | 0
  Dead | 1 | 2 | 1 | 3

7. Primary Outcome: Cumulative Dose of FE 202158
Description: Cumulative dose of FE 202158 was calculated from Day 1 up to Day 7.
Time Frame: as for outcome 1
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Measure: Mean (60% Confidence Interval); unit: ng/kg
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 5 | 13
ng/kg
  Day 1 (Post 12 h) | 2451 [2226.3 to 2675.8] | 3276.3 [2941.3 to 3611.3] | 2946 [2426.2 to 3465.8] | 2377 [2220.2 to 2533.7]
  Day 1 (Post 24 h) | 4217.4 [3736.5 to 4698.3] | 5502.2 [4698.7 to 6305.7] | 4927.3 [4064.8 to 5789.8] | 3818.8 [3429.6 to 4208.0]
  Day 2 (Post 36 h) | 4463.9 [3877.0 to 5050.7] | 7535.9 [6206.2 to 8865.7] | 5842 [4554.6 to 7129.4] | 4619.2 [4005.0 to 5233.4]
  Day 2 (Post 48 h) | 4523.9 [3900.8 to 5146.9] | 9185 [7405.2 to 10963.9] | 6716 [4674.3 to 8757.6] | 5225 [4401.7 to 6048.3]
  Day 3 (Post 72 h) | 4523.9 [3900.8 to 5146.9] | 11511.4 [9096.1 to 13926.7] | 7902 [4758.8 to 11045.1] | 5860.1 [4763.9 to 6956.4]
  Day 4 (Post 96 h) | 4523.9 [3900.8 to 5146.9] | 12204.6 [9365.7 to 15043.4] | 7999.8 [4765.3 to 11234.3] | 6298.6 [4939.5 to 7657.7]
  Day 5 (Post 120 h) | 4523.9 [3900.8 to 5146.9] | 12865.3 [9561.7 to 16168.9] | 7999.8 [4765.3 to 11234.3] | 6621.8 [5033.5 to 8210.1]
  Day 6 (Post 144 h) | 4523.9 [3900.8 to 5146.9] | 13543.7 [9724.0 to 17363.3] | 7999.8 [4765.3 to 11234.3] | 6696.5 [5052.9 to 8340.1]
  Day 7 (Post 168 h) | 4523.9 [3900.8 to 5146.9] | 13543.7 [9724.0 to 17363.3] | 7999.8 [4765.3 to 11234.3] | 7003.7 [5126.0 to 8881.5]

8. Primary Outcome: Infusion Rate of FE 202158
Description: Infusion rate of FE 202158 was presented from Day 1 up to Day 7.
Time Frame: as for outcome 1
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Measure: Mean (Standard Deviation); unit: ng/kg/min
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 5 | 13
ng/kg/min
  Day 1 (Post 12 h) | 3.25 (1.29) | 4.13 (2.09) | 3.08 (2.56) | 2.43 (1.41)
  Day 1 (Post 24 h) | 0.94 (1.88) | 3.39 (2.37) | 1.59 (2.19) | 1.39 (1.65)
  Day 2 (Post 36 h) | 0.23 (0.47) | 2.66 (2.27) | 2.08 (2.77) | 1.25 (1.76)
  Day 2 (Post 48 h) | 0.00 (0.00) | 2.51 (2.29) | 1.79 (3.57) | 0.69 (1.28)
  Day 3 (Post 72 h) | 0.00 (0.00) | 0.82 (2.02) | 0.61 (1.22) | 0.39 (1.08)
  Day 4 (Post 96 h) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.33 (1.08)
  Day 5 (Post 120 h) | 0.00 (0.00) | 0.99 (2.21) | 0.00 (0.00) | 0.00 (0.00)
  Day 6 (Post 144 h) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 7 (Post 168 h) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.33 (1.08)

9. Primary Outcome: Cumulative Dose of Norepinephrine
Description: Norepinephrine was infused as required to maintain the target mean arterial pressure, if the highest infusion rate allowed of experimental drug FE 202158 did not provide adequate vasopressor support. Cumulative dose of norepinephrine was calculated from Day 1 up to Day 7.
Time Frame: as for outcome 1
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed. One patient in the 7.5 ng/kg/min group started the vasopressor support without prior administration of norepinephrine, and MAP was adequately controlled as needed.
Measure: Mean (60% Confidence Interval); unit: µg/kg
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 4 | 13
µg/kg
  Day 1 (Post 12 h) | 358.1 [91.8 to 624.3] | 172.1 [96.5 to 247.8] | 118.0 [12.7 to 223.3] | 73.1 [47.2 to 99.0]
  Day 1 (Post 24 h) | 720.8 [131.8 to 1309.7] | 338.0 [171.5 to 504.6] | 357.5 [17.8 to 697.2] | 149.5 [90.4 to 208.6]
  Day 2 (Post 36 h) | 720.8 [131.8 to 1309.7] | 406.2 [214.7 to 597.6] | 778.2 [26.9 to 1529.5] | 197.8 [111.4 to 284.2]
  Day 2 (Post 48 h) | 720.8 [131.8 to 1309.7] | 495.5 [296.4 to 694.5] | 778.4 [27.2 to 1529.7] | 232.8 [120.6 to 345.1]
  Day 3 (Post 72 h) | 720.8 [131.8 to 1309.7] | 669.0 [390.8 to 947.2] | 778.4 [27.2 to 1529.7] | 279.1 [129.5 to 428.7]
  Day 4 (Post 96 h) | 720.8 [131.8 to 1309.7] | 829.6 [438.1 to 1221.1] | 778.4 [27.2 to 1529.7] | 303.1 [133.6 to 472.6]
  Day 5 (Post 120 h) | 720.8 [131.8 to 1309.7] | 1039.5 [473.7 to 1605.2] | 778.4 [27.2 to 1529.7] | 307.8 [134.4 to 481.2]
  Day 6 (Post 144 h) | 720.8 [131.8 to 1309.7] | 1152.0 [489.2 to 1814.7] | 778.4 [27.2 to 1529.7] | 307.8 [134.4 to 481.2]
  Day 7 (Post 168 h) | 720.8 [131.8 to 1309.7] | 1152.0 [489.2 to 1814.7] | 778.4 [27.2 to 1529.7] | 311.1 [134.9 to 487.2]

10. Primary Outcome: Infusion Rate of Norepinephrine
Description: Norepinephrine was infused as required to maintain the target mean arterial pressure, if the highest infusion rate allowed of experimental drug FE 202158 did not provide adequate vasopressor support. Infusion rates and all changes in infusion rates of norepinephrine were recorded continuously during the 7 day maximum treatment period.
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: µg/kg/min
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 4 | 13
µg/kg/min
  Day 1 (Post 12 h) | 0.341 (0.691) | 0.281 (0.444) | 0.215 (0.405) | 0.111 (0.197)
  Day 1 (Post 24 h) | 0.010 (0.020) | 0.222 (0.402) | 0.639 (1.280) | 0.089 (0.188)
  Day 2 (Post 36 h) | 0.000 (0.000) | 0.049 (0.101) | 0.000 (0.000) | 0.061 (0.171)
  Day 2 (Post 48 h) | 0.000 (0.000) | 0.105 (0.215) | 0.004 (0.008) | 0.057 (0.188)
  Day 3 (Post 72 h) | 0.000 (0.000) | 0.120 (0.270) | 0.000 (0.000) | 0.024 (0.079)
  Day 4 (Post 96 h) | 0.000 (0.000) | 0.184 (0.411) | 0.000 (0.000) | 0.005 (0.016)
  Day 5 (Post 120 h) | 0.000 (0.000) | 0.172 (0.385) | 0.000 (0.000) | 0.000 (0.000)
  Day 6 (144 h) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  Day 7 (Post 168 h) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.006 (0.021)

11. Primary Outcome: Time to Septic Shock Resolution
Description: The Kaplan-Meyer estimation of time to out of septic shock was estimated where time to (first) septic shock resolution was defined as time of end of infusion regimen. Intermittent off treatment periods were regarded as part of the shock duration.
  Time to all but one patient out of septic shock is presented.
Time Frame: Day 1 up to Day 28
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Measure: Number; unit: Hours
Groups:
- Full Analysis Set: The full analysis data set (FAS) comprised data from all dosed patients.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 30
Hours
  3.75 ng/kg/min (n=5) | 23
  5.0 ng/kg/min (n=7) | 75
  7.5 ng/kg/min (n=5) | 37
  Modified 3.75 ng/kg/min (n=13) | 89

12. Secondary Outcome: Mortality
Description: Collection of data on mortality was performed on Day 28 in addition to the collection of data on time of stay in intensive care unit and hospital.
Time Frame: Day 1 up to Day 28
Population: Full analysis set (FAS) was the primary dataset of interest. FAS comprised of all patients who were dosed.
Measure: Number; unit: patients
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 5 | 13
patients
  Alive | 4 | 3 | 4 | 10
  Dead | 1 | 2 | 1 | 3

13. Secondary Outcome: Adverse Effects on Lab Parameters, Vital Signs and Electrocardiogram
Description: Significant changes for vital signs (blood pressure, heart rate, mean arterial pressure), electrocardiogram (ECG), and laboratory parameters (clinical chemistry, haematology, haemostasis, and urinary parameters).
Time Frame: Day 1 up to Day 7, and at follow-up assessments performed 24-72 hours after end of IMP infusion
Population: The safety analysis set comprised of all allocated and dosed patients and were analyzed according to the actual dosing regimen received.
Measure: Number; unit: patients
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min
Number analyzed (Participants) | 5 | 7 | 5 | 13
patients
  Patients with adverse effects on lab parameters | 0 | 0 | 0 | 0
  Patients with adverse effects on vital signs | 0 | 0 | 0 | 0
  Patients with adverse effects on electrocardiogram | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from start of study up to the end of trial on Day 28, or end of follow-up period as applicable.
Description: Collection of adverse events comprised the patient's positive response to questions about their health, symptoms spontaneously reported by the patient, and clinically relevant changes and abnormalities observed by the investigator.
Groups:
- Total: Summation of adverse events in all treatment arms
Arm/Group | Infusion Regimen 1: 3.75 ng/kg/Min | Infusion Regimen 2: 5.0 ng/kg/Min | Infusion Regimen 3: 7.5 ng/kg/Min | Infusion Regimen 4: Modified 3.75 ng/kg/Min | Total
Serious Adverse Events (participants affected / at risk) | 1/5 | 4/7 | 2/5 | 3/13 | 10/30
Other Adverse Events (participants affected / at risk) | 4/5 | 7/7 | 4/5 | 12/13 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infusion Regimen 1: 3.75 ng/kg/Min (N=5) | Infusion Regimen 2: 5.0 ng/kg/Min (N=7) | Infusion Regimen 3: 7.5 ng/kg/Min (N=5) | Infusion Regimen 4: Modified 3.75 ng/kg/Min (N=13) | Total (N=30)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Intestinal ischemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic congestion (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colostomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Distributive shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infusion Regimen 1: 3.75 ng/kg/Min (N=5) | Infusion Regimen 2: 5.0 ng/kg/Min (N=7) | Infusion Regimen 3: 7.5 ng/kg/Min (N=5) | Infusion Regimen 4: Modified 3.75 ng/kg/Min (N=13) | Total (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocardial depression (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cytolytic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic congestion (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 5 (5)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats in this trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.